CLINICAL TRIAL: NCT06269328
Title: Evaluatıon The Effects Of Anesthesıcs And Surgıcal Treatment On Sleep Qualıty In Patıents That Posterıor Spınal Instrumentatıon Plannıng
Brief Title: Measuring Sleep Quality In Patients That Posterior Spinal Instrumentatıon Plannıng
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Elifgül Ulutaş, Specialist, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011-KAEK-26/463
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2022-07

CONDITIONS: Sleep Disorder; Sleep, Inadequate; Total ıntravenous Anesthesia; Inhalation Anesthesia
Keywords: Anesthesia; General anesthesia; Sleep quality; Total ıntravenous anesthesia; Inhalation anesthesia
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Deprivation; Sleep Initiation and Maintenance Disorders | interventions — Propofol; Remifentanil; Anesthesia, Inhalation; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA group (Active Comparator): Patients will be anesthetized with total ıntravenous anesthesia by propofol and remifentanyl infusion. End of the procedure all patients will be extubated and awakened in the operating room. İntravenous morphine patient-controlled analgesia will be used in the postoperative period.
  Interventions: Other: Total ıntravenous anesthesia with propofol and remifentanil for anesthetic maintenance
- İnhalation group (Active Comparator): Patients will be anesthetized with induction of propofol and sevoflurane (inhalational agent) will be used for maintenance. End of the procedure all patients will be extubated and awakened in the operating room. İntravenous morphine patient-controlled analgesia will be used in the postoperative period.
  Interventions: Other: Inhalation anesthesia with sevoflurane for anesthetic maintenance

INTERVENTIONS:
Other: Total ıntravenous anesthesia with propofol and remifentanil for anesthetic maintenance — For anesthesia induction, intravenous propofol was used at doses of 1-2 mg/kg, fentanyl at 2mcg/kg, lidocaine at 1mg/kg, and rocuronium at doses of 1mg/kg. After then anesthesia maintained with propofol iv 75-100 µg kg-1 min-1 and remifentanyl iv 0.05-0.2 µg kg-1 min-1 infusion.
  Arms: TIVA group
Other: Inhalation anesthesia with sevoflurane for anesthetic maintenance — For anesthesia induction, intravenous propofol was used at doses of 1-2 mg/kg, fentanyl at 2mcg/kg, lidocaine at 1mg/kg, and rocuronium at doses of 1mg/kg. After then anesthesia was maintained with inhalation anesthetic (50% O2/Air with Sevoflurane 2% )
  Arms: İnhalation group

SUMMARY:
Postoperative sleep disorders have serious problems with cognition, pain perception, sustained circadian rhythm, psychomotor function, metabolic function, catabolic responses, and continuity. The relationship between general anesthesia and sleep disturbances following surgery is still unclear. Since the risk of sleep disorders after surgery is high, it is important to determine the efficiency of the interval with automatic sleep disorders. By evaluating how major orthopedic surgery and general anesthesia applied to posterior spinal instrumentation divides sleep quality, risk management allows determining the factors involved in the peroperative period and thus facilitating surgical results and patient comfort.

DETAILED DESCRIPTION:
Sleep is one of the basic physiological needs of humans. It is necessary for the mind to perform functions such as learning, memory and cognition. Sleep disorders, which can occur for short or long periods in the perioperative period, affect many patients. Studies have shown that approximately 8.8-79.1% of patients experience perioperative sleep disorders, and this situation can continue for a long time after surgery.

According to animal and human studies, anesthetic agents may cause sleep disorders in the postoperative period. Anesthetics can disrupt the normal sleep-wake cycle and thus cause insomnia and poor sleep quality. Since postoperative pain and emotional changes will also cause sleep disturbances, the view that general anesthesia impairs postoperative sleep quality has not yet been proven.

Different types of surgery have varying effects on sleep quality. Patients state that they experience more sleep disruption due to pain, especially after orthopedic surgery. Patients' sleep quality may be even worse due to the greater trauma caused by major surgery. Thoracolumbar posterior instrumentation is a frequently used method in the treatment of spinal instability resulting from spinal trauma, neoplasia, congenital or degenerative diseases. Therefore, we wanted to specifically evaluate this patient group in our study.

Old age, female gender and chronic diseases are among the factors that increase the likelihood of experiencing sleep disorders. Environmental factors and healthcare practices in the hospital may contribute to sleep disturbances. Postoperative environment change, inadequate beds, noise and lights in the ward, medical staff, night treatment and nursing controls, machine noises, postoperative diets and warnings from the urinary catheter are additional factors that affect patients' sleep.

Evaluation of sleep disorders is mainly based on clinical symptoms (difficulty falling asleep, early awakening, night terrors, nightmares or abnormal behavior during the sleep period) and auxiliary objective scales. Subjective sleep quality assessment mainly scales: Pittsburgh Sleep Quality Index questionnaire (PSQI), Pittsburgh Insomnia Rating Scale (PIRS), Insomnia Severity Index (ISI), Athens Insomnia Scale, Epworth Sleepiness Scale (ESS), General Sleep Disturbance Scale (GSDS). The most commonly used assessment in clinical studies is the PSQI. PSQI has high reliability and validity, but evaluates over a one-month period. The PIRS_20 scale, which is a self-assessment survey, is a scale created by the Department of Psychiatry at the University of Pittsburgh and evaluates the sleep quality of participants in the last week. It generally consists of a questionnaire with a total of twenty items, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, and sleep disorders. Scoring ranges from 0 to 60. A score of 20 and above indicates poor sleep quality, while as the score increases, sleep quality deteriorates.

Sleep disorders can negatively impact patient recovery, contributing to higher rates of postoperative complications such as neurological and cardiovascular morbidity and delayed postoperative recovery. They are also risk factors for cardiovascular and cerebrovascular diseases such as myocardial infarction, as well as dementia, obesity, diabetes, hypertension, depression, pain and even death. It is also considered an important risk factor for the development of delirium. Despite posing a significant threat to public health, sleep disorders remain poorly understood, underdiagnosed, and poorly managed, especially in perioperative patients. The potential negative consequences of sleep disorders indicate the need for greater attention to this issue.

Despite its importance, sleep quality assessment is not a part of the routine preoperative evaluation of patients and does not receive enough attention. Peroperative sleep assessment can provide information for anesthesiologists and surgeons that may allow early interventions. There are no guidelines or sufficient number of studies for clinical use.

In this study, PIRS-20 (Pittsburg Insomnia Rating Scale_20), VAS (Visual Analog Scale), State Anxiety Scale (STAI-1) will be used. In addition, the Oswestry Functional Disability Scale, SRS-22 (Scoliosis Research Society-22) questionnaire, EQ-5D-5L General Quality of Life Scale, SF-36 Quality of Life Scale, which are routinely used in orthopedic clinics, are used to evaluate anesthesia and surgery in patients undergoing posterior spinal instrumentation. The investigators aimed to evaluate changes in sleep patterns caused by trauma and simultaneously anxiety and pain levels.

The aim of this research is to evaluate how major orthopedic surgery and general anesthesia affect the sleep quality of patients who underwent posterior spinal instrumentation.

The primary hypothesis of this study is that total intravenous anesthesia with propofol and remifentanil is superior to inhalation anesthesia with sevoflurane in terms of sleep quality. In this process, the investigators aimed to identify risk factors for patients, thus improving surgical results and patient comfort.

ELIGIBILITY:
Inclusion criteria:

* Elective total hip arthroplasty planning
* 18 years and older patients
* ASA score between I-III
* Approved and signed the informed consent form

Exclusion Criteria:

* Patients under 18 years of age
* Patients with ASA score 4 and above
* Patients who do not accept informed consent
* Those who refuse to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Subjective sleep quality (evaluated by PIRS-20 (Pitssburg Insomnia Rating Scale) | Preoperative status a month before surgery and a day before surgery and one week postoperatively]
  Sleep quality evaluated by PIRS-20 (Pitssburg Insomnia Rating Scale) , a scale provides ranging from 0 to 60 , with a high score indicating a poor quality of sleeping.

SECONDARY OUTCOMES:
Subjective anxiety level | Preoperative status a month before surgery and a day before surgery and one week postoperatively]
  Anxiety level evaluated by STAI (The State Trait Anxiety Inventory), a scale provides ranging from 20 to 80, with a high score indicating high levels of anxiety.
Subjective pain level | Preoperative status a month before surgery and a day before surgery and one week postoperatively]
  Pain level evaluated by VAS (Visuel analog scale) , a scale provides ranging from 0 to 10, with a high score indicating high levels of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Elifgül Ulutaş, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No